CLINICAL TRIAL: NCT05462834
Title: Impact of Nocturnal Hypoxemia on Glucose in High Altitude Sleep Disordered Breathing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in foreign component policy at NIH.
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); PRISMA A.B. (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00329264; K23HL155730 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sleep-Disordered Breathing; Glucose Intolerance
MeSH Terms: conditions — Sleep Apnea Syndromes; Glucose Intolerance | interventions — Compressed Air

STUDY DESIGN:
Intervention Model Description: 2 intervention periods lasting 14 days, separated by a 7-day washout
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressed Air then Supplemental Oxygen (Experimental)
  Interventions: Other: Compressed Air; Other: Supplemental Oxygen
- Supplemental Oxygen then Compressed Air (Experimental)
  Interventions: Other: Compressed Air; Other: Supplemental Oxygen

INTERVENTIONS:
Other: Compressed Air — Participants will be instructed to use compressed air during sleep as a placebo control.
Other: Supplemental Oxygen — Participants will be instructed to use supplemental oxygen at rate of 2lpm during sleep.

SUMMARY:
Sleep disordered breathing is associated with impaired glucose tolerance and incident diabetes. Nocturnal hypoxemia is a potential stimulus of glucose intolerance. It is especially severe and highly prevalent in high altitude residents. Intervening on nocturnal hypoxemia may therefore improve glucose control and decrease the public health burden in high altitude populations.

The objective of this study is to examine the impact of hypoxemia on glucose homeostasis in high altitude residents. The investigators will address this objective by examining the effect of supplemental oxygen on glucose in a randomized cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents of Puno, Peru

Exclusion Criteria:

* Recent travel to low altitude (<3000 m)
* Oxygen use
* Pregnancy
* Morbid obesity (BMI > 40 kg/m2)
* Current smoking
* Diabetes
* Other sleep disorders (e.g. circadian rhythm disorder or insomnia)
* Use of open fires in the home (i.e. for cooking or heat)
* Chronic Mountain Sickness (CMS) as defined by a daytime oxyhemoglobin saturation < 85%, Qinghai CMS >10 or excessive erythrocytosis as defined by hemoglobin >19 g/dL in women or >21 g/dL in men.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Mean glucose level | 14 days after start of intervention
  average glucose (mg/dL) during sleep assessed via continuous glucose monitoring

SECONDARY OUTCOMES:
Mean fasting glucose level | 14 days after start of intervention
  Mean fasting glucose level (mg/dL)
Mean fasting insulin | 14 days after start of intervention
  Fasting insulin (U/mL)
Morning blood pressure | 14 days after start of intervention
  Morning blood pressure (mmHg)
Inflammatory marker interleukin-6 (IL-6) | 14 days after start of intervention
  Inflammatory marker interleukin-6 (IL-6) (pg/mL) level in plasma assessed by electrochemiluminescence as a measure of systemic inflammation
Tumor Necrosis Factor alpha (TNF-a) level in blood (picogram/milliliter) | 14 days after start of intervention
  Tumor Necrosis Factor alpha level in blood as a marker of inflammation
C-Reactive Protein (CRP) level in blood (mg/L) | 14 days after start of intervention
  C-Reactive Protein (CRP) level in blood as a marker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Luu Pham, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No